CLINICAL TRIAL: NCT02048995
Title: Neural and Visual Responses to Light in Bipolar Disorder: A Novel Putative Biomarker
Acronym: LightEyeBD
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Dorothy Sit, Associate Professor of Psychiatry and Behavioral Sciences, Northwestern University
Other Study IDs: PRO14010387
Record Dates: First submitted 2014-01-24; First posted 2014-01-29 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Bipolar Depression
Keywords: Bipolar Disorder; Depression; Light Therapy; Contrast Sensitivity; Visual Evoked Potential; Visual or Neural Responses; Biomarker
MeSH Terms: conditions — Bipolar Disorder; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Bipolar Depressed: Bipolar Depressed - are participants with Bipolar Disorder Type I or II and a current episode of major depression which is confirmed on the SCID interview
- Healthy Comparator: Healthy Comparator - are participants without mental disorders, alcohol or substance disorders confirmed by the SCID-interview

SUMMARY:
Objective. Bipolar Disorders (BD) are a major public health problem. The investigators still lack knowledge of the mechanisms which contribute to BD. Hence treatments are few and limited, and clinical decision making is less refined. Currently, the investigators are investigating the effects of midday bright light therapy for the treatment of bipolar depression (University of Pittsburgh IRB approved protocol titled Light Therapy for Bipolar Disorder, IRB#: PRO09020546). In this study, the investigators propose to investigate a possible biological mechanism which might explain response to light treatment in depressed bipolar patients.

DETAILED DESCRIPTION:
The study goal is to understand how the response to light therapy relates to changes in vision, brain function and improvement in bipolar symptoms. The aims are to investigate mood levels plus the eye and brain responses to visual contrast stimuli in healthy comparators (HC) and bipolar depressed patients.

Study Design and Methods. Overview. The investigators plan to enroll 18-50 year old adults with BD Type I or II and a current episode of major depression on stable-dosed antimanic drugs, and age and sex-matched HC - without mental disorders. Depressed patients with BD will be assigned randomly to receive active light therapy vs inactive comparator for 6 weeks. The investigators will examine responses to contrast stimuli from measures of visual evoked potentials and electro-retinography in HC and depressed bipolar patients before and after 6-weeks of daily midday light therapy. The investigators will assess repeated measures of mood symptom levels, attention and circadian rhythms.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-50 years.
* DSM-IV BD Type I or II, current major depressive episode
* Stable-dosed antidepressant drug for 4 weeks or more only with concurrent antimanic drug.
* Controlled thyroid disease.
* Subjects with preexisting eye diseases will be included specific exceptions are described in the Exclusion Criteria.
* Able to provide informed consent.
* Stable minimum dose of antimanic drug for 4weeks or more.
* Stable unchanged psychotherapy for 16 weeks or more.
* Permitted drugs for sleep at low doses.

Exclusion Criteria:

* Certain specific eye diseases (retinal disease, untreated cataracts or macular degeneration)
* Photosensitizing drugs such as phenothiazines (chlorpromazine), antimalarial drugs, melatonin and hypericum.
* Acute psychosis (DSM-IV Criteria)
* Rapid cycling in the past 1 year
* Alcohol or substance abuse or dependence in the past 6 months.
* Current symptoms of hypomania or mania i.e. ManiaRatingScale=5
* Recent history of a suicide attempt (3 months) or active suicidal ideation (SIGH-ADS item H11=2 or more)
* Treatment with propranolol (Inderal), exogenous melatonin, chronic NSAIDS.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: community patient sample
Sampling Method: Probability Sample
Enrollment: 91 (Estimated)
Dates: Start 2014-02; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
visual evoked potentials (VEP) waveforms (mean amplitudes or latencies) | Week 0 and Week 6
  Visual Evoked Potential (VEP). This is a test which is used to assess visual cortical responses. The VEP recordings will be assessed at different contrast levels (80%, 16% and 7%) for the patient groups (BD vs HC). To assess the change in visual cortical responses, we will compare differences in the VEP responses between Weeks 0 and 6 between the groups.
Electroretinography (ERG) waveforms (mean amplitudes or latencies) | Week 0 and Week 6
  Electroretinogram (ERG). This is a test which is used to assess electrical responses of the retina. The ERG recordings will be assessed at different contrast levels (80%, 16% and 7%) for the patient groups (BD vs HC). To assess the change in retinal responses, we will compare differences in ERG responses between Weeks 0 and 6 between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Sit, M.D., Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States